CLINICAL TRIAL: NCT04483999
Title: Turkish Validity and Reliability Study of Virtual Reality Sickness Questionnaire
Status: Completed | Type: Observational
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, HATİCE ÇETİN, Research Assisstant, Hacettepe University
Other Study IDs: VRSQ9
Record Dates: First submitted 2020-07-20; First posted 2020-07-23 (Actual); Last update posted 2023-04-18 (Actual); Status verified 2023-04

CONDITIONS: Sickness Behavior
Keywords: virtual reality; sickness; validity; reliability; turkish
MeSH Terms: conditions — Illness Behavior

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study is planned for the cultural adaptation and validity of the "Virtual Reality Sickness Questionnaire".

DETAILED DESCRIPTION:
Virtual reality (SG) creates a virtual environment that reflects a real environment and offers various experiences to users. Motion sickness can be observed in people after using virtual reality applications or simulation devices in education. There are questionnaires in the literature such as "Simulator Sickness Questionnaire" and "Motion Sickness Questionnaire". However, these questionnaires are specific surveys to evaluate symptoms that develop after vehicle handling or use of simulation devices for pilot training, while they are not ideal questionnaires to evaluate symptoms that may develop after virtual reality applications. Because there are important differences between virtual reality systems and simulation systems in terms of the appearance of motion disturbance symptoms. For this reason, "Virtual Reality Sickness Questionnaire" has been developed that can evaluate these symptoms.

There is no Turkish version of the "Virtual Reality Sickness Questionnaire" in the literature. For this reason, this study is planned for the cultural adaptation and validity of the "Virtual Reality Sickness Questionnaire".

ELIGIBILITY:
Inclusion Criteria:

* Not having mental - cognitive problems,
* Being a volunteer

Exclusion Criteria:

* Oculomotor and vestibular disease
* Cardiovascular, neurological and gastrointestinal problems

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy people
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2021-06-30 (Actual); Primary Completion 2023-01-30 (Actual); Study Completion 2023-03-30 (Actual)

PRIMARY OUTCOMES:
Virtual Reality Sickness Questionnaire | Change from Baseline sickness after 1 hour later.
  This questionnaire assess virtual reality sickness. This questionnaire consists of 2 subtitles as oculomotor and disorientation. It contains 9 symptoms in total. Each symptom is scored between 0 and 3 with the Likert type scoring system. Each subtitle adapted to be calculated by dividing the total score to a score system in itself like person receives%. The total score of the questionnaire will be obtained by averaging the total scores of the two subtitles.
graybiel scale | Change from Baseline sickness after 1 hour later.
  This questionnaire assess virtual reality sickness. Total score ranges from 0-50. 0-2 points are interpreted as "light susceptibility to motion sickness", 3-7 points as "moderate susceptibility to motion sickness", 8-15 points as "extreme susceptibility to motion sickness", and values above 16 are "Definitive motion sickness".

SECONDARY OUTCOMES:
international physical activity questionnaire | All of the participants will assess at baseline with this scale.
  This questionnaire assess physical activity level. The physical activity levels are classified as (< 600 MET-min/week), which is the physically inactive level (level I); (600-3000 METmin/week), which is the level in medium-level (level II) and (> 3000 MET-min/week), which is the high physical activity level.
tampa kinesiophobia scale | All of the participants will assess at baseline with this scale.
  This questionnaire assess kinesiophobia. The four-point Likert scoring is used in this scale (1 = I do not agree at all, 4 = I agree completely). The total score is calculated after reversing the items 4, 8, 12 and 16. Scoring ranges between 17 and 68 with the higher scores indicating higher levels of kinesiophobia perception.

CONTACTS AND LOCATIONS:
Overall Officials: NEZİRE KOSE, Principal Investigator — Hacettepe University
Locations (1):
- Hatice Çetin, Ankara, Sıhhiye, Turkey (Türkiye)

REFERENCES:
- [Background] Kim HK, Park J, Choi Y, Choe M. Virtual reality sickness questionnaire (VRSQ): Motion sickness measurement index in a virtual reality environment. Appl Ergon. 2018 May;69:66-73. doi: 10.1016/j.apergo.2017.12.016. Epub 2018 Jan 16. PMID 29477332
- See also: URL — https://pubmed.ncbi.nlm.nih.gov/29477332/